CLINICAL TRIAL: NCT01099358
Title: Phase 2 Study to Evaluate the Pharmacokinetics and Drug-Drug Interaction of Cetuximab and Cisplatin in Patients With Advanced Solid Tumors
Brief Title: Study in Advanced Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13418; I4E-MC-JXBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-30; First posted 2010-04-07 (Estimated); Results first posted 2016-12-13 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Solid Tumor
Keywords: Cancer of Head; Cancer of Head and Neck; Cancer of Neck; Cancer of the Head; Cancer of the Head and Neck; Cancer of the Neck; Head and Neck Cancer; Head Cancer; Head Neoplasms; Head, Neck Neoplasms; Neck Cancer; Neck Neoplasms; Solid Neoplasm; Carcinoma; Sarcoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma; Sarcoma | interventions — Cetuximab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cetuximab and Cisplatin (D) (Experimental): Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m²) cetuximab administered (admin) intravenously (I.V) on week 1, day 1.
  100 mg/m² cisplatin administered I.V on week 1, day 1. Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/m²/day (d) administered starting on week 1, day 1.
  After 1 cycle, participants may continue treatment as determined by the physician until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: 5 - Fluorouracil
- Cetuximab and Cisplatin (C) (Experimental): Cycle 1 (4 weeks, combination therapy):
  100 mg/m² Cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 400 mg/m² cetuximab admin I.V on week 2, day 1. 250 mg/m² cetuximab admin I.V on week 3 and 4, day 1.
  Cycle 2-6 (3 weeks combination therapy):
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 250 mg/m² cetuximab admin I.V on week 1, 2, and 3, day 1.
  After 6 cycles, participants may then receive weekly cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and cisplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: 5 - Fluorouracil
- Cetuximab on Cisplatin (B) (Experimental): Cycle 1:
  400 mg/m² cetuximab admin I.V on week 1, day 1. 250 mg/m² cetuximab admin I.V on week 2 and 3, day 1.
  Cycle 2:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1- 4.
  250 mg/m² cetuximab admin I.V on week 1-3, day 1.
  Cycle 3 + :
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  250 mg/m² cetuximab admin I.V on week 1-3, day 1.
  After 6 cycles, participants may then receive weekly cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and cisplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: 5 - Fluorouracil
- Cisplatin on Cetuximab (A) (Experimental): Cycle 1:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  400 mg/m² cetuximab admin I.V on week 2, day 1. 250 mg/m² cetuximab admin I.V on week 3, day 1.
  Cycle 2 +:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  250 mg/m² cetuximab admin I.V on weeks 1-3, day 1.
  After 7 cycles, participants may then receive weekly Cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and cisplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Drug: 5 - Fluorouracil

INTERVENTIONS:
Drug: Cetuximab — Administered Intravenously
Drug: Cisplatin — Administered Intravenously
Drug: 5 - Fluorouracil — Administered Intravenously

SUMMARY:
The primary purpose of this study is to help answer the following research question(s):

* To see how the body absorbs, processes, and gets rid of cetuximab when the drug is taken in combination with cisplatin [pharmacokinetic (PK) analysis]
* To see if any drug interactions occur between cetuximab and cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically advanced solid tumor that is resistant to standard therapy or for which there is no standard therapy.
* The participant has measurable or non-measurable disease.
* The participant has a life expectancy of greater than 3 months.
* The participant has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* The participant has adequate hematologic function as defined by absolute neutrophil count greater than or equal to 1500/microliter (μL), hemoglobin greater than or equal to 9 grams/deciliter (g/dL), and platelet count greater than or equal to 100,000/μL.
* The participant has adequate hepatic function as defined by a total bilirubin less than or equal to 2 x the upper limit of normal (ULN), aspartate transaminase (AST, SGOT) and alanine transaminase (ALT, SGPT) less than or equal to 3 x the ULN (or less than or equal to 5 x the ULN in the presence of known liver metastases).
* The participant has adequate renal function as defined by serum creatinine less than or equal to 1.5 x the institutional ULN or creatinine clearance greater than or equal to 60 mL/min for participants with creatinine levels above the ULN.
* The participant has the ability to understand, and the willingness to sign, a written informed consent document.
* If the participant has received prior therapy with platinum, the time to the first treatment of study drug from the last platinum exposure is >28 days.

Exclusion Criteria:

* The participant has symptomatic brain or leptomeningeal metastasis.
* The participant has not recovered from Adverse Events due to agents administered more than 4 weeks earlier. Neurotoxicity, if present, must have improved to Grade less than 2 per the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v 3.0.
* The participant is receiving any other investigational agent(s).
* The participant is receiving concurrent treatment with other anticancer therapy, including chemotherapy, immunotherapy, hormonal therapy, radiation therapy (RT), chemoembolization, or targeted therapy. Participants receiving palliative radiation therapy to bony metastases prior to the first dose of study medication are eligible.
* The participant is receiving therapy with immunosuppressive agents.
* The participant has known drug or alcohol abuse.
* The participant has uncontrolled hypertension defined as systolic blood pressure greater than or equal to 180 millimeters of mercury (mm Hg) or diastolic blood pressure greater than or equal to 130 mm Hg.
* The participant has a history of allergic reactions attributed to compounds of chemical or biologic composition similar to those of cetuximab or cisplatin.
* The participant has a medical or psychological condition that would not permit the participant to complete the study or sign informed consent.
* The participant has clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency.
* The participant, if female, is pregnant (confirmed by serum or urine beta-human chorionic gonadotropin [β-HCG] pregnancy test) or breastfeeding
* The participant has had a known positive test result for the human immunodeficiency virus.
* The participant has an active infection (requiring intravenous [IV] antibiotics), including tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-04; Primary Completion 2015-10 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (5):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Kansas Medical Center, Fairway, Kansas
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - University of North Carolina, Chapel Hill, North Carolina
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas
- Canada (2):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to protocol amendment in September 2011,any newly enrolled participants were placed into cetuximab and cisplatin(C) arm only.After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab(cet) and cisplatin(D) arm only. Group(Grp)A (cisplatin [cis]) completed 3 infusions(inf) of cet (Weeks(wk) 2,3, & 4
Pre-assignment Details: [wk 4 = wk 1 of cycle(cyc) 2]) & 2 inf of cis(wk 1 & 4) first 4 wks.Grp B (cet) completed 4 inf of cet (wk 1-4) & 1 inf of cis(wk 4) first 4 wks. Grp C(cis and cet) completed 4 inf of cet(wk 2,3,4, & 5) & 2 inf of cis(wk 1 & 5) first 5 wk. Grp D(cis) completed 1 inf of cet(cyc 1) & 1 inf of cis(wk 1 of cyc 1) and without deviation.
Period: Overall Study
Arm/Group | Cisplatin on Cetuximab (A) | Cetuximab on Cisplatin (B) | Cetuximab and Cisplatin (C) | Cetuximab and Cisplatin (D)
Started | 4 | 6 | 21 | 16
Received at Least One Dose of Study Drug | 3 | 6 | 20 | 15
Completed | 1 | 5 | 13 | 12
Not Completed | 3 | 1 | 8 | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants (All Participants (Group A, B, C and D): A:Cycle1:100mg/m² cisplatin(cs) I.V on week(w)1,day(d)1. 5-FU as a 96-hour(h) C.I. of 1000 mg/m²/d starting (st) on w 1,d 1-4.
  400mg/m² cetuximab(ct) I.V on w 2,d 1.250mg/m² ct I.V on w 3,d 1.Cycle 2+100mg/m² cs I.V on w 1,d 1.5-FU as a 96-h C.I. of 1000mg/m²/d st on w 1,d 1-4.250mg/m² ct I.V on w 1-3,d 1.
  B:Cycle1:400mg/m² ct I.V on w 1,d 1.250mg/m² ct I.V on w 2&3,d 1.Cycle 2:100mg/m² cs I.V on w 1, d 1.5-FU as a 96-h C.I. of 1000mg/m²/d st on w 1,d 1- 4.250mg/m² ct I.V on w 1-3,d 1.Cycle 3 +:100mg/m² cs I.V on w 1,d 1.5-FU as a 96-h C.I. of 1000mg/m²/d st on w 1,d 1-4.
  250mg/m² ct I.V on w 1-3,d 1. C:Cycle1:100mg/m² cs I.V on w 1, d 1. 5-FU as a 96-h C.I. of 1000mg/m²/d st on w 1,d 1.400 mg/m² ct I.V on w 2,d 1.250mg/m² ct I.V on w 3&4,d 1.Cycle2-6:100mg/m² cs I.V on w 1,d 1.5-FU as a 96-h C.I. of 1000mg/m²/d st w 1,d 1. 250mg/m² ct I.V w 1,2,&3,d 1.
  D:Cycle1:400mg/m² ct I.V w 1,d 1.100mg/m² cs I.V w 1,d 1.Optional 5-FU as a 96-h C.I. of 1000mg/m²/d st w 1,d 1.
Arm/Group | All Participants (All Participants (Group A, B, C and D)
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (11.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 34
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Canada | 16
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Total Cisplatin Pharmacokinetics (PK): Area Under the Concentration (AUC) Versus Time Curve From Time Zero to Infinity (AUC[0-∞])
Time Frame: Groups A and C: Cycle 1,Day 1 and Cycle 2 Day 1; Baseline (Prior to Cisplatin Infusion), 1, 1.50, 2, 3, 5, 8, 24, 72 hours (After the Start of Cisplatin Infusion).
Population: All participants who received at least one dose of study drug who were enrolled in Group A or C and had evaluable PK data. Study design by intent did not collect data from Group B or Group D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliters (μg*h/mL)
Groups:
- Cetuximab (A and C); Cetuximab and Cisplatin (A and C): Cisplatin on Cetuximab (A)
  Cycle 1:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  400 mg/m² cetuximab admin I.V on week 2, day 1. 250 mg/m² cetuximab admin I.V on week 3, day 1.
  Cycle 2 +:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  250 mg/m² cetuximab admin I.V on weeks 1-3, day 1.
  Cetuximab and Cisplatin (C)
  Cycle 1 (4 weeks, combination therapy):
  100 mg/m² Cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 400 mg/m² cetuximab admin I.V on week 2, day 1. 250 mg/m² cetuximab admin I.V on week 3 and 4, day 1.
  Cycle 2-6 (3 weeks combination therapy):
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 250 mg/m² cetuximab admin I.V on week 1, 2, and 3, day 1.
Arm/Group | Cetuximab (A and C) | Cetuximab and Cisplatin (A and C)
Number analyzed (Participants) | 5 | 5
micrograms*hour/milliliters (μg*h/mL) | 324 (24.5) | 338 (26.1)

2. Primary Outcome: Cetuximab Pharmacokinetics: Area Under the Concentration Versus Time Curve During One Dosing Interval at Steady State (AUC τ,ss)
Time Frame: Group B:Cycle 1,Day 15 and Cycle 2, Day 1 and Group C: Cycle 1, Day 22 and Cycle 2, Day 1: Baseline (Prior to Cetuximab Infusion),1, 2, 4, 8, 24, 72, 120, and 168 hours (After the Start of Cetuximab Infusion).
Population: All participants who received at least one dose of study drug who were enrolled in Group B or C and had evaluable PK data. Study design by intent did not collect data from Group A or Group D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour/milliliters (μg*h/mL)
Groups:
- Cetuximab (B and C); Cetuximab and Cisplatin (B and C): Cetuximab on Cisplatin (B) Cycle 1:400 mg/m² cetuximab admin I.V on week 1, day 1. 250 mg/m² cetuximab admin I.V on week 2 and 3, day 1.
  Cycle 2:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5-FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1- 4.
  250 mg/m² cetuximab admin I.V on week 1-3, day 1.
  Cycle 3 + :
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5-FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  250 mg/m² cetuximab admin I.V on week 1-3, day 1.
  Cetuximab and Cisplatin (C) Cycle 1 100 mg/m² cisplatin admin I.V on week 1, day 1. 5-FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 400 mg/m² cetuximab admin I.V on week 2, day 1. 250 mg/m² cetuximab admin I.V on week 3 and 4, day 1.
  Cycle 2-6 100 mg/m² cisplatin admin I.V on week 1, day 1. 5-FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 250 mg/m² cetuximab admin I.V on week 1, 2, and 3, day 1.
Arm/Group | Cetuximab (B and C) | Cetuximab and Cisplatin (B and C)
Number analyzed (Participants) | 14 | 14
micrograms*hour/milliliters (μg*h/mL) | 15000 (25.7) | 16200 (22.5)

3. Primary Outcome: Total Cisplatin Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliters(μg/mL)
Arm/Group | Cetuximab (A and C) | Cetuximab and Cisplatin (A and C)
Number analyzed (Participants) | 5 | 5
micrograms/milliliters(μg/mL) | 4.08 (23.2) | 4.22 (10.2)

4. Primary Outcome: Cetuximab Pharmacokinetics: Maximum Observed Plasma Concentration at Steady State (Cmax,ss)
Time Frame: as for outcome 2
Population: All participants who received at least one dose of study drug who were enrolled in Group B and C and had evaluable PK data. Study design by intent did not collect data from Group A or Group D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (μg/mL)
Arm/Group | Cetuximab (B and C) | Cetuximab and Cisplatin (B and C)
Number analyzed (Participants) | 14 | 14
micrograms per milliliters (μg/mL) | 194 (20.6) | 192 (12.8)

5. Primary Outcome: Total Cisplatin Pharmacokinetics: Measurement of the Time After Administration When the Maximum Plasma Concentration is Reached (Tmax)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Cetuximab (A and C) | Cetuximab and Cisplatin (A and C)
Number analyzed (Participants) | 5 | 5
Hours (h) | 1.02 [0.97 to 1.50] | 1.05 [1.00 to 1.42]

6. Primary Outcome: Cetuximab Pharmacokinetics: Measurement of the Time After Administration When the Maximum Plasma Concentration is Reached (Tmax)
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Cetuximab (B and C) | Cetuximab and Cisplatin (B and C)
Number analyzed (Participants) | 14 | 14
Hours (h) | 2.00 [1.00 to 4.05] | 1.99 [1.00 to 4.18]

7. Primary Outcome: Cetuximab Pharmacokinetics: Confirmatory Serum Concentration
Time Frame: Group D:Cycle 1, Day 1: Prior to Cisplatin Infusion.
Population: All participants who received at least one dose of study drug who were enrolled in Group D and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliters (μg/mL)
Groups:
- Cetuximab (D): Cetuximab and Cisplatin (D)
  Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m²) cetuximab administered (admin) intravenously (I.V) on week 1, day 1.
  100 mg/m² cisplatin administered I.V on week 1, day 1. Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/m²/day (d) administered starting on week 1, day 1.
Arm/Group | Cetuximab (D)
Number analyzed (Participants) | 11
micrograms per milliliters (μg/mL) | 198 (18.5)

ADVERSE EVENTS:
Description: All participants who received at least one dose of study drug.
Groups:
- Cisplatin on Cetuximab (A): Cisplatin on Cetuximab (A)
  Cycle 1:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  400 mg/m² cetuximab admin I.V on week 2, day 1. 250 mg/m² cetuximab admin I.V on week 3, day 1.
  Cycle 2 +:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  250 mg/m² cetuximab admin I.V on weeks 1-3, day 1.
  After 7 cycles, participants may then receive weekly Cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and cisplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
- Cetuximab on Cisplatin (B): Cetuximab on Cisplatin (B)
  Cycle 1:
  400 mg/m² cetuximab admin I.V on week 1, day 1. 250 mg/m² cetuximab admin I.V on week 2 and 3, day 1.
  Cycle 2:
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1- 4.
  250 mg/m² cetuximab admin I.V on week 1-3, day 1.
  Cycle 3 + :
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1-4.
  250 mg/m² cetuximab admin I.V on week 1-3, day 1.
  After 6 cycles, participants may then receive weekly cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and cisplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
- Cetuximab and Cisplatin (C): Cetuximab and Cisplatin (C)
  Cycle 1 (4 weeks, combination therapy):
  100 mg/m² Cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 400 mg/m² cetuximab admin I.V on week 2, day 1. 250 mg/m² cetuximab admin I.V on week 3 and 4, day 1.
  Cycle 2-6 (3 weeks combination therapy):
  100 mg/m² cisplatin admin I.V on week 1, day 1. 5- FU admin as a 96-hour C.I. of 1000 mg/m²/d admin starting on week 1, day 1. 250 mg/m² cetuximab admin I.V on week 1, 2, and 3, day 1.
  After 6 cycles, participants may then receive weekly cetuximab monotherapy until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  Due to protocol amendment in September 2011, any newly enrolled participants were placed into cetuximab and cisplatin (C) arm only. After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
- Cetuximab and Cisplatin (D): Cetuximab and Cisplatin (D)
  Cycle 1 (1 week, combination therapy):
  400 milligrams per square meter (mg/m²) cetuximab administered (admin) intravenously (I.V) on week 1, day 1.
  100 mg/m² cisplatin administered I.V on week 1, day 1. Optional 5- fluorouracil (FU) administered as a 96-hour continuous infusion (C.I.) of 1000 mg/m²/day (d) administered starting on week 1, day 1.
  After 1 cycle, participants may continue treatment as determined by the physician until progression of disease, unacceptable toxicity, or another withdrawal criterion is met.
  After protocol amendment February 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.
Arm/Group | Cisplatin on Cetuximab (A) | Cetuximab on Cisplatin (B) | Cetuximab and Cisplatin (C) | Cetuximab and Cisplatin (D)
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/6 | 12/20 | 6/15
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 20/20 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin on Cetuximab (A) (N=3) | Cetuximab on Cisplatin (B) (N=6) | Cetuximab and Cisplatin (C) (N=20) | Cetuximab and Cisplatin (D) (N=15)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin on Cetuximab (A) (N=3) | Cetuximab on Cisplatin (B) (N=6) | Cetuximab and Cisplatin (C) (N=20) | Cetuximab and Cisplatin (D) (N=15)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (8) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (10) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 6 (13) | 3 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 7 (7) | 4 (4)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 9 (14) | 9 (11)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (6) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (3) | 18 (25) | 8 (10)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 9 (14) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (2) | 8 (13) | 4 (6)
Asthenia (General disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (4) | 3 (4) | 10 (18) | 7 (7)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 2 (3) | 7 (12) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 2 (6) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 6 (19) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 1 (3) | 5 (6) | 1 (2)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 4 (5) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 3 (9) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 1 (4) | 7 (11) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (6) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 2 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 6 (13) | 3 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (5) | 1 (3) | 12 (32) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 5 (9) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (6) | 10 (19) | 8 (10)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (3) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (6) | 3 (3)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to protocol amendment in Sep 2011,any newly enrolled participants were placed into cetuximab and cisplatin (C) arm only. After protocol amendment June 2014, any newly enrolled participants will be placed into cetuximab and cisplatin (D) arm only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days